CLINICAL TRIAL: NCT00559650
Title: Placebo Controlled, Randomized, Double-blind, Multi-center, Multinational Phase IIb Study to Investigate the Efficacy and Tolerability of BAY58-2667 Given Intravenously in Patients With Decompensated Chronic Congestive Heart Failure
Brief Title: Placebo Controlled, Randomized, Double-blind, Multi-center Study to Investigate the Efficacy and Tolerability of BAY58-2667
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12480; 2007-003059-36 (EudraCT Number)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Congestive Heart Failure
Keywords: Acute decompensated heart failure; Double blind study,; BAY58-2667; Soluble guanylate cyclase activator
MeSH Terms: conditions — Heart Failure | interventions — BAY 58-2667

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)

INTERVENTIONS:
Drug: Placebo — Will be standard therapy and placebo versus, Uptitration from 100-600µg/g, intravenous, over maximum 48 hours
  Arms: Arm 1
Drug: Cinaciguat (BAY58-2667) — Will be standard therapy and BAY 58-2667, Uptitration from 100-600µg/g, intravenous, over maximum 48 hours
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess a dose titration scheme, of a new drug (BAY58-2667) given intravenously, to evaluate if this is safe and can help to improve the well-being, symptoms (e.g. breathing) and outcome of decompensated heart failure. Patients living with chronic heart failure have a risk of increased number of hospitalisations because of worsening of their condition (decompensated heart failure). The current treatment of acute heart failure consists of oxygen and medical treatment with vasodilators and positive inotropic agents (drugs, which should strengthen the pump function of the heart) which have their limitations. Therefore there is a need for new drugs in treatment of acute heat failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with decompensated chronic congestive heart failure, NYHA functional class III-IV, either ischemic or non-ischemic, requiring hospitalization, and with clinical indication for parenteral pharmacotherapy and invasive hemodynamic monitoring (i.e indwelling Swan-Ganz pulmonary artery catheter) and PCWP >/= 18 mmHg.
* Patients must have the clinical diagnosis of CHF made at least 3 month prior to enrollment.
* Male or female patients, age 18 years or more.

Exclusion Criteria:

* Females of child-bearing potential.
* Acute de-novo heart failure.
* Acute myocardial infarction and/or myocardial infarction within 30 days.
* Valvular heart disease requiring surgical intervention during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome measure will be the change of pulmonary capillary wedge pressure (PCWP) from baseline to 8 hours versus placebo. | 8 hours

SECONDARY OUTCOMES:
Quality of Life | Up to 30 days Follow-up
Rehospitalization | Up to 30 days Follow-up
Other hemodynamic measurements | Up to 48 hours
  Right atrial pressure (RAP); mean pulmonary artery pressure (PAP mean); pulmonary artery systolic pressure (PASP); pulmonary artery diastolic pressure (PADP); cardiac output (CO); cardiac index (CI); mean arterial pressure (MAP); pulmonary vascular resistance (PVR); pulmonary vascular resistance index (PVRI); systemic vascular resistance (SVR); and systemic vascular resistance index (SVRI）
Safety variables | Up to 30 days follow up
  Treatment-emergent adverse events, laboratory parameters, renal function, in-hospital mortality, length of stay at intensive care unit, and 30-day mortality / morbidity.
Plasma concentrations | During both the titration and maintenance phases were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (67):
- United States (6):
  - San Diego, California
  - Washington D.C., District of Columbia
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Dallas, Texas
- Canada (3):
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Ste-Foy, Quebec
- Croatia (2):
  - Split
  - Zagreb
- Czechia (4):
  - Brno
  - Hradec Králové
  - Pilsen
  - Prague
- Estonia (2):
  - Tallinn
  - Tartu
- Germany (12):
  - Heidelberg, Baden-Wurttemberg
  - Würzburg, Bavaria
  - Bad Nauheim, Hesse
  - Greifswald, Mecklenburg-Vorpommern
  - Bad Oeynhausen, North Rhine-Westphalia
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Halle, Saxony-Anhalt
  - Berlin, State of Berlin
  - Erfurt, Thuringia
  - Jena, Thuringia
- Hungary (4):
  - Budapest
  - Debrecen
  - Vác
  - Zalaegerszeg
- Israel (4):
  - Haifa, Israel
  - Jerusalem
  - Ramat Gan
  - Safed
- Italy (6):
  - Bologna, Emilia-Romagna
  - Ferrara, Emilia-Romagna
  - Milan, Lombardy
  - Pavia, Lombardy
  - Perugia, Umbria
  - Bergamo
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (5):
  - Gdansk
  - Krakow
  - Szczecin
  - Wroclaw
  - Zabrze
- Moscow, Russia
- Serbia (2):
  - Belgrade
  - Kamenitz
- Slovenia (4):
  - Celje
  - Golnik
  - Ljubljana
  - Murska Sobota
- Spain (5):
  - Santiago de Compostela, A Coruña
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Girona, Girona
  - Majadahonda, Madrid
- Sweden (2):
  - Gothenburg
  - Uppsala
- United Kingdom (3):
  - Chesterfield, Derbyshire
  - Barnet, Hertfordshire
  - Harrow, Middlesex

REFERENCES:
- [Result] Erdmann E, Semigran MJ, Nieminen MS, Gheorghiade M, Agrawal R, Mitrovic V, Mebazaa A. Cinaciguat, a soluble guanylate cyclase activator, unloads the heart but also causes hypotension in acute decompensated heart failure. Eur Heart J. 2013 Jan;34(1):57-67. doi: 10.1093/eurheartj/ehs196. Epub 2012 Jul 9. PMID 22778174
- See also: Click here and search for Bayer product information provided by EMA — http://www.clinicaltrialsregister.eu